CLINICAL TRIAL: NCT05705544
Title: Robotic Versus Electromagnetic Bronchoscopy for Pulmonary LesIon AssessmeNT: (the RELIANT Trial)
Acronym: RELIANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Fabien Maldonado, Professor of Medicine and Thoracic Surgery, MD, MSc, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 221255
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Pulmonary Lesions
Keywords: Electromagnetic navigational bronchoscopy; Shape-sensing catheter bronchoscopy; Diagnostic yield

STUDY DESIGN:
Intervention Model Description: This study will be performed as a pragmatic, cluster randomized controlled trial with parallel group assignment.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: It is not possible to blind the bronchoscopist or the patient to the platform used for each procedure, as they are both large distinctive-appearing pieces of equipment.
  However, thoracic pathologists (the outcomes assessor) and bronchoscopy schedulers (the care provider team) will remain blinded, such that allocations should be unable to influence their histopathological interpretation or scheduling of procedures in a given OR, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ILLUMISITE™ Platform (EMN bronchoscopy) (Active Comparator): Participants in the ILLUMISITE™ Platform arm will undergo a diagnostic bronchoscopy with the ILLUMISITE™ Platform (EMN) machine.
  Interventions: Device: ILLUMISITE™ Platform (EMN bronchoscopy)
- Ion™ Endoluminal System (SSCB bronchoscopy) (Active Comparator): Participants in the Ion™ Endoluminal System arm will undergo a diagnostic bronchoscopy with the Ion™ Endoluminal System (SSCB) machine.
  Interventions: Device: Ion™ Endoluminal System (SSCB bronchoscopy)

INTERVENTIONS:
Device: ILLUMISITE™ Platform (EMN bronchoscopy) — Providers will utilize the ILLUMISITE™ Platform (EMN) machine to perform a diagnostic bronchoscopy procedure.
  Arms: ILLUMISITE™ Platform (EMN bronchoscopy)
Device: Ion™ Endoluminal System (SSCB bronchoscopy) — Providers will utilize the Ion™ Endoluminal System (SSCB) machine to perform a diagnostic bronchoscopy procedure.
  Arms: Ion™ Endoluminal System (SSCB bronchoscopy)

SUMMARY:
This is an investigator-initiated, cluster randomized controlled trial. The primary objective is to compare the diagnostic yield of the Ion™ Endoluminal System (SSCB) to the ILLUMISITE™ Platform (EMN bronchoscopy) in patients undergoing bronchoscopy for peripheral pulmonary lesion (PPL) evaluation.

DETAILED DESCRIPTION:
Peripheral pulmonary lesions (PPLs) are often biopsied to assess for the presence of infection, inflammation, or malignancy. Tissue can be acquired in a variety of ways: surgical resection, percutaneous transthoracic needle biopsy, or bronchoscopic biopsy. Bronchoscopy is commonly pursued to determine PPL etiology, with over 500,000 performed annually in the US alone. Advanced imaging and navigational guidance systems are required to accurately approach small peripheral lesions bronchoscopically. A variety of navigational technologies are currently available, including electromagnetic navigational bronchoscopy (EMN), virtual bronchoscopy, thin and ultrathin bronchoscopes, and endobronchial ultrasound. No comparative data exist regarding the relative performance of these competing technologies, which are all considered standard of care and currently used interchangeably based on personal preferences and availability.

EMN platforms dominate the current navigational bronchoscopy market. The largest prospective multicenter study assessing EMN performance showed a diagnostic yield of 73%. The more recent addition of intraprocedural digital tomosynthesis has been reported to increase EMN diagnostic yield to 75-83%; this feature is included in the ILLUMISITE™ electromagnetic navigational bronchoscopy platform (Medtronic, Minneapolis, MN, U.S.) and is labeled "fluoroscopic navigation".

Recently, the FDA cleared a novel navigational technology: shape-sensing catheter bronchoscopy (SSCB), via the 510(k) pathway. This pathway requires a technical demonstration of safety and efficacy similar to that of an existing predicate device but does not usually require clinical data. Since market release in 2019, single-center prospective cohort data have emerged suggesting SSCB diagnostic yield is comparable to EMN, but no high-quality comparative data exist regarding the relative performance of these two technologies. Despite this important knowledge/data gap, SSCB has become a popular platform in the advanced bronchoscopist community. High-quality comparative data are required to inform optimal patient care. Additionally, EMN and SSCB platforms are considered capital purchases, each costing hundreds of thousands of dollars. Hence, it is also important for health care systems to have high quality data as they consider device purchases. VUMC currently utilizes both SSCB and EMN and they are used interchangeably in our two operating rooms. Patients are typically assigned arbitrarily to procedures using either platform based on operating room availability.

Thus, the investigator proposes a randomized controlled study to test the hypothesis that the diagnostic yield of SSCB is not inferior to EMN in patients undergoing bronchoscopy to biopsy a PPL.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older at time of bronchoscopy.

Scheduled for navigational bronchoscopy for the evaluation of a peripheral pulmonary lesion.

Exclusion Criteria:

Enrolled in a different study requiring use of one of these specific platforms (i.e., ILLUMISITE™ Platform (EMN) or Ion™ Endoluminal System (SSCB)).

Subject declines to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Maldonado, MD, MSc, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available (including data dictionaries) after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years.
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.

REFERENCES:
- [Background] Criner GJ, Eberhardt R, Fernandez-Bussy S, Gompelmann D, Maldonado F, Patel N, Shah PL, Slebos DJ, Valipour A, Wahidi MM, Weir M, Herth FJ. Interventional Bronchoscopy. Am J Respir Crit Care Med. 2020 Jul 1;202(1):29-50. doi: 10.1164/rccm.201907-1292SO. PMID 32023078
- [Background] Cicenia J, Avasarala SK, Gildea TR. Navigational bronchoscopy: a guide through history, current use, and developing technology. J Thorac Dis. 2020 Jun;12(6):3263-3271. doi: 10.21037/jtd-2019-ndt-11. PMID 32642249
- [Background] Folch EE, Pritchett MA, Nead MA, Bowling MR, Murgu SD, Krimsky WS, Murillo BA, LeMense GP, Minnich DJ, Bansal S, Ellis BQ, Mahajan AK, Gildea TR, Bechara RI, Sztejman E, Flandes J, Rickman OB, Benzaquen S, Hogarth DK, Linden PA, Wahidi MM, Mattingley JS, Hood KL, Lin H, Wolvers JJ, Khandhar SJ; NAVIGATE Study Investigators. Electromagnetic Navigation Bronchoscopy for Peripheral Pulmonary Lesions: One-Year Results of the Prospective, Multicenter NAVIGATE Study. J Thorac Oncol. 2019 Mar;14(3):445-458. doi: 10.1016/j.jtho.2018.11.013. Epub 2018 Nov 23. PMID 30476574
- [Background] Katsis J, Roller L, Aboudara M, Pannu J, Chen H, Johnson J, Lentz RJ, Rickman O, Maldonado F. Diagnostic Yield of Digital Tomosynthesis-assisted Navigational Bronchoscopy for Indeterminate Lung Nodules. J Bronchology Interv Pulmonol. 2021 Oct 1;28(4):255-261. doi: 10.1097/LBR.0000000000000766. PMID 33734149
- [Background] Aboudara M, Roller L, Rickman O, Lentz RJ, Pannu J, Chen H, Maldonado F. Improved diagnostic yield for lung nodules with digital tomosynthesis-corrected navigational bronchoscopy: Initial experience with a novel adjunct. Respirology. 2020 Feb;25(2):206-213. doi: 10.1111/resp.13609. Epub 2019 Jul 2. PMID 31265204
- [Background] Avasarala SK, Roller L, Katsis J, Chen H, Lentz RJ, Rickman OB, Maldonado F. Sight Unseen: Diagnostic Yield and Safety Outcomes of a Novel Multimodality Navigation Bronchoscopy Platform with Real-Time Target Acquisition. Respiration. 2022;101(2):166-173. doi: 10.1159/000518009. Epub 2021 Sep 3. PMID 34515222
- [Background] Agrawal A, Hogarth DK, Murgu S. Robotic bronchoscopy for pulmonary lesions: a review of existing technologies and clinical data. J Thorac Dis. 2020 Jun;12(6):3279-3286. doi: 10.21037/jtd.2020.03.35. PMID 32642251
- [Background] Kalchiem-Dekel O, Connolly JG, Lin IH, Husta BC, Adusumilli PS, Beattie JA, Buonocore DJ, Dycoco J, Fuentes P, Jones DR, Lee RP, Park BJ, Rocco G, Chawla M, Bott MJ. Shape-Sensing Robotic-Assisted Bronchoscopy in the Diagnosis of Pulmonary Parenchymal Lesions. Chest. 2022 Feb;161(2):572-582. doi: 10.1016/j.chest.2021.07.2169. Epub 2021 Aug 9. PMID 34384789
- [Derived] Chen SC, Chen H, Paez R, Gatto CL, Lentz RJ, Maldonado F. A randomization strategy for a cluster-randomized controlled trial with variable operating room availability. Contemp Clin Trials. 2025 Oct;157:108057. doi: 10.1016/j.cct.2025.108057. Epub 2025 Aug 28. PMID 40885487
- [Derived] Paez R, Lentz RJ, Duke JD, Siemann JK, Salmon C, Dahlberg GJ, Ratwani AP, Casey JD, Chen H, Chen SC, Shojaee S, Rickman OB, Gatto CL, Rice TW, Maldonado F. Robotic versus Electromagnetic Bronchoscopy for Peripheral Pulmonary Lesions: A Randomized Trial (RELIANT). Am J Respir Crit Care Med. 2025 Sep;211(9):1644-1651. doi: 10.1164/rccm.202409-1846OC. PMID 40460390
- [Derived] Paez R, Lentz RJ, Salmon C, Siemann JK, Low SW, Casey JD, Chen H, Chen SC, Avasarala S, Shojaee S, Rickman OB, Lindsell CJ, Gatto CL, Rice TW, Maldonado F; Vanderbilt Learning Healthcare System Platform Investigators. Robotic versus Electromagnetic bronchoscopy for pulmonary LesIon AssessmeNT: the RELIANT pragmatic randomized trial. Trials. 2024 Jan 19;25(1):66. doi: 10.1186/s13063-023-07863-3. PMID 38243291
- [Derived] Paez R, Lentz RJ, Salmon C, Siemann JK, Low SW, Casey JD, Chen H, Chen SC, Avasarala S, Shojaee S, Rickman OB, Lindsell CJ, Gatto CL, Rice TW, Maldonado F. Robotic versus Electromagnetic Bronchoscopy for Pulmonary LesIon AssessmeNT: the RELIANT pragmatic randomized trial. Res Sq [Preprint]. 2023 Aug 28:rs.3.rs-3222369. doi: 10.21203/rs.3.rs-3222369/v1. PMID 37693467
- See also: U.S. Food and Drug Administration. 510(K) Clearances. Accessed November 5, 2021 — https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ILLUMISITE™ Platform (EMN Bronchoscopy) | Ion™ Endoluminal System (SSCB Bronchoscopy)
Started | 208 | 203
Completed | 208 | 203
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ILLUMISITE™ Platform (EMN Bronchoscopy): Participants in the Electromagnetic navigational bronchoscopy (ENB) arm underwent a diagnostic bronchoscopy with the ILLUMISITE™ Platform (EMN) machine.
  ILLUMISITE™ Platform (EMN bronchoscopy): Providers utilized the ILLUMISITE™ Platform (EMN) machine to perform a diagnostic bronchoscopy procedure.
- Ion™ Endoluminal System (SSCB Bronchoscopy): Participants in the Robotic assisted bronchoscopy (RAB) arm underwent a diagnostic bronchoscopy with the Ion™ Endoluminal System (SSCB) machine.
  Ion™ Endoluminal System (SSCB bronchoscopy): Providers utilized the Ion™ Endoluminal System (SSCB) machine to perform a diagnostic bronchoscopy procedure.
- Total: Total of all reporting groups
Arm/Group | ILLUMISITE™ Platform (EMN Bronchoscopy) | Ion™ Endoluminal System (SSCB Bronchoscopy) | Total
Number analyzed (Participants) | 208 | 203 | 411
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.0 [59.0 to 75.0] | 69.0 [61.0 to 74.0] | 67.0 [60.0 to 74.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 101 | 201
  Male | 108 | 102 | 210
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 189 | 188 | 377
  Race: Black or African American | 15 | 15 | 30
  Race: Asian | 3 | 0 | 3
  Race: Unknown or unable to report | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Non-Hispanic | 202 | 198 | 400
  Ethnicity: Hispanic | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 208 | 203 | 411
Current malignancy [Count of Participants; unit: Participants] | 42 | 51 | 93
Prior malignancy [Count of Participants; unit: Participants] | 73 | 71 | 144
Body Mass Index, median [Median (Inter-Quartile Range); unit: Kg/m^2] | 26.8 [23.9 to 30.4] | 26.5 [23.0 to 30.6] | 26.6 [23.4 to 30.5]
Anticoagulation or antiplatelet [Count of Participants; unit: Participants] | 85 | 86 | 171
Smoking history [Count of Participants; unit: Participants]
  Current | 44 | 44 | 88
  Former | 94 | 97 | 191
  Never | 70 | 62 | 132
Lesion size, largest diameter (mm), median [Median (Inter-Quartile Range); unit: mm] | 20.0 [14.0 to 29.0] | 18.0 [12.0 to 28.0] | 19.0 [13.0 to 28.0]
Lesion location (outer 1/3 of the chest) [Count of Participants; unit: Participants] | 141 | 139 | 280
Lesion density (solid) [Count of Participants; unit: Participants] | 176 | 171 | 347
Lesion spiculation [Count of Participants; unit: Participants] | 41 | 62 | 103
Bronchus sign present [Count of Participants; unit: Participants] | 128 | 112 | 240
Lesion distance from pleura (mm), median [Median (Inter-Quartile Range); unit: mm] | 4.0 [0.0 to 14.0] | 6.0 [0.0 to 18.0] | 5.0 [0.0 to 15.5]

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Yield
Description: Diagnostic yield is defined as the proportion of procedures that results in acquisition of lesional tissue. Lesional tissue is defined by the presence of histopathological findings that readily explain the presence of a pulmonary lesion.
  The following common histopathological findings are pre-specified as lesional:
  i. Malignant ii. "Specific benign" findings accounting for the presence of a PPL
  1. organizing pneumonia, or
  2. frank purulence/robust neutrophilic inflammation, or
  3. granulomatous inflammation, or
  4. other specific benign finding findings such as hamartoma, amyloidoma or other uncommon causes of PPLs with distinctive pathological patterns.
Time Frame: 7 days post-enrollment
Measure: Count of Participants; unit: Participants
Groups:
- ILLUMISITE™ Platform (EMN Bronchoscopy): Participants in the Electromagnetic navigational bronchoscopy (ENB) arm will undergo a diagnostic bronchoscopy with the ILLUMISITE™ Platform (EMN) machine.
  ILLUMISITE™ Platform (EMN bronchoscopy): Providers will utilize the ILLUMISITE™ Platform (EMN) machine to perform a diagnostic bronchoscopy procedure.
- Ion™ Endoluminal System (SSCB Bronchoscopy): Participants in the Robotic assisted bronchoscopy (RAB) arm will undergo a diagnostic bronchoscopy with the Ion™ Endoluminal System (SSCB) machine.
  Ion™ Endoluminal System (SSCB bronchoscopy): Providers will utilize the Ion™ Endoluminal System (SSCB) machine to perform a diagnostic bronchoscopy procedure.
Arm/Group | ILLUMISITE™ Platform (EMN Bronchoscopy) | Ion™ Endoluminal System (SSCB Bronchoscopy)
Number analyzed (Participants) | 208 | 203
Participants | 157 | 158

2. Secondary Outcome: Duration of Procedure
Description: Defined as time from the start of airway registration to the removal of the bronchoscope after completion of navigation procedures
Time Frame: Duration of procedure, approximately 60 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | ILLUMISITE™ Platform (EMN Bronchoscopy) | Ion™ Endoluminal System (SSCB Bronchoscopy)
Number analyzed (Participants) | 208 | 203
minutes | 32.0 [25.0 to 43.3] | 37.0 [29.0 to 48.0]

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | ILLUMISITE™ Platform (EMN Bronchoscopy) | Ion™ Endoluminal System (SSCB Bronchoscopy)
All-Cause Mortality (participants affected / at risk) | 0/208 | 0/203
Serious Adverse Events (participants affected / at risk) | 7/208 | 5/203
Other Adverse Events (participants affected / at risk) | 5/208 | 0/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ILLUMISITE™ Platform (EMN Bronchoscopy) (N=208) | Ion™ Endoluminal System (SSCB Bronchoscopy) (N=203)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Anesthesia Complication (Injury, poisoning and procedural complications) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ILLUMISITE™ Platform (EMN Bronchoscopy) (N=208) | Ion™ Endoluminal System (SSCB Bronchoscopy) (N=203)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Persistent dyspnea post-procedure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Persistent Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT05705544/Prot_001.pdf
  • Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT05705544/SAP_002.pdf
  • Informed Consent Form (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/44/NCT05705544/ICF_000.pdf